CLINICAL TRIAL: NCT02786628
Title: Assessing Physical Fitness in Cancer Patients With Cardiopulmonary Exercise Testing and Wearable Data Generation
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC 1543
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Malignant Solid Tumour; Hematologic Malignancies; Planned Hematopoietic Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Exercise Test; Patient Generated Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Solid tumor malignancies: 15 patients. Will participate in physical performance testing and patient-generated health data.
  Interventions: Other: Physical performance testing and patient-generated health data
- Hematologic malignancies: 15 patients. Will participate in physical performance testing and patient-generated health data.
  Interventions: Other: Physical performance testing and patient-generated health data
- Hematopoietic cell transplantation: 15 patients. Will participate in physical performance testing and patient-generated health data.
  Interventions: Other: Physical performance testing and patient-generated health data

INTERVENTIONS:
Other: Physical performance testing and patient-generated health data — All patients will complete cardiopulmonary exercise testing and 6 minute walk distance performance testing prior to a cycle of chemotherapy (or transplant) and wear a Fitbit Charge HR for the duration of one cycle of chemotherapy.

SUMMARY:
The primary objective of this study is to assess the feasibility of a multi-institutional study that collects cardiopulmonary exercise testing and 6 minute walk distance performance testing prior to a cycle of chemotherapy (or transplant), followed by collection of patient generated health data (wearable activity monitors and patient reported outcomes) for the subsequent month. In addition to demonstrating feasibility, the study looks to generate preliminary data that supports the capacity of physical performance testing and patient-generated health data to complement clinician-rated performance status in patients receiving chemotherapy.

DETAILED DESCRIPTION:
Physical fitness, based on tests of physical performance and measurements of daily activity, can serve as both a risk stratification variable and clinical outcome for patients prior to or during cytotoxic chemotherapy. Many cytotoxic therapies cause premature aging and frailty in a sizable portion of patients, so measuring and improving physical function may also limit late morbidity and mortality in certain patient populations. Clinician-rated performance status (cPS; e.g., ECOG or Karnofsky PS) in addition to organ-specific function have been used to prognosticate risk and determine treatment strategy, but cPS only readily identifies individuals with significant functional compromise. Objective evaluations of physical function, such as aerobic capacity and measured daily activity, may have greater potential to improve the precision of performance status evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumor or hematologic malignancies who are planning to receive a cycle of cytotoxic chemotherapy or patients who are planning to receive stem cell transplant.
* Age ≥ 18
* At least 6 weeks out from surgical resection
* Presence of working email address
* Access to internet at home and access to electronic device(s) capable of charging and syncing the Fitbit
* Ability to read and understand English
* Ability to understand and comply with study procedures including wearing Fitbit for the entire length of the study
* Approval of attending oncologist for participation in the study
* Hb ≥ 8 g/dL (most recent lab draw)
* Willingness and ability to provide written informed consent

Exclusion Criteria:

* Dementia, altered mental status, or psychiatric condition that would prohibit the understanding or rendering of informed consent
* Presence of cardiac disease including acute MI within past 6 weeks, unstable angina, uncontrolled arrhythmias causing symptoms, active endocarditis, myocarditis, or pericarditis,symptomatic aortic stenosis, uncontrolled heart failure, syncope in the past 6 weeks, severe untreated hypertension at rest (>180 mmHg systolic, >100 mmHg diastolic)
* Acute pulmonary embolism or thrombosis of lower extremities in the past 6 weeks
* Uncontrolled asthma
* Pulmonary edema
* Suspected dissecting aneurysm
* Room air desaturation at rest </= 88%
* Respiratory failure
* Acute noncardiopulmonary disorder that may be aggravated by exercise
* Mental impairment leading to inability to cooperate with instructions
* Orthopedic impairment that compromises exercise performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 patients with cancer undergoing a cycle of cytotoxic chemotherapy or bone marrow transplant.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients being approached that agree to participate in the study | 7 months
  This is measure 1 for determining study feasibility
Proportion of enrolled patients who complete CPET and 6MWD test without significant testing-related adverse events | 7 months
  This is measure 2 for determining study feasibility
Proportion of recruited patients who wear Fitbit for at least 8 hours per day | 7 months
  This is measure 3 for determining study feasibility
Proportion of patients for whom all data is successfully recorded within database | 7 months
  This is measure 4 for determining study feasibility; using UNC PRO-Core and Fitabase to collect information

SECONDARY OUTCOMES:
Compare pre-treatment aerobic capacity (VO2max or 6MWD) with post-treatment average measured steps per day | 7 months
  Comparison made to determine if pre-treatment aerobic capacity is predictive of post-treatment steps per day.
Compare pre-treatment clinician-rated performance status and aerobic capacity (VO2max or 6MWD) with post-treatment average steps per day | 7 months
  Comparison made to determine which pre-treatment value better predicts post-treatment steps per days.
Compare pre-treatment aerobic capacity (VO2max or 6MWD) and post-treatment average measured steps per day among the three cohorts (solid tumor, hematologic malignancies, hematopoietic cell transplantation) | 7 months
Compare average measured steps per day and patient-reported symptomatic toxicities | 7 months
Compare resting heart rate trajectories (as measured by Fitbit) before and after chemotherapy | 7 months
Compare resting heart rates as measured from VO2max testing with resting heart rates as measured by Fitbit | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Grover, MD, Principal Investigator — University of North Carolina, Chapel Hill; William A Wood, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wood WA, Dilip D, Derkach A, Grover NS, Elemento O, Levine R, Thanarajasingam G, Batsis JA, Bailey C, Kannappan A, Devine SM, Artz AS, Ligibel JA, Basch E, Kent E, Glass J. Wearable sensor-based performance status assessment in cancer: A pilot multicenter study from the Alliance for Clinical Trials in Oncology (A19_Pilot2). PLOS Digit Health. 2023 Jan 26;2(1):e0000178. doi: 10.1371/journal.pdig.0000178. eCollection 2023 Jan. PMID 36812616